CLINICAL TRIAL: NCT04847115
Title: Treatment of Fifth Metatarsal Zone 3 Fractures - A Prospective, Randomized, Controlled Trial
Brief Title: Treatment of Fifth Metatarsal Zone 3 Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201144
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Fractures, Stress; Metatarsal Fracture
MeSH Terms: conditions — Fractures, Stress | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: Prospecitve, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative (Active Comparator): The patients in this arm will be treated operatively with intramedullar screw osteosynthesis. In addition to this, they will weight bear as tolareted in a walking boot orthosis for six weeks.
  Interventions: Procedure: Operative; Other: Walking boot orthosis
- Non-operative (Active Comparator): The patients in this arm will have non-operative treatment with a walking boot orthosis for six weeks. They will weight bear as tolerated
  Interventions: Other: Walking boot orthosis

INTERVENTIONS:
Procedure: Operative — Intramedullary screw fixation
  Other Names: Osteosynthesis
  Arms: Operative
Other: Walking boot orthosis — Non-operative treatment with walking boot orthosis for six weeks. The non-operative study arm will use walking boot orthosis only. The operative study arm will use walking boot orthosis as adjuvant treatment.

SUMMARY:
The fifth metatarsal is one of the bones where stress fractures can occur. Current literature provides support for both operative and non-operative treatment, but is mostly based on retrospective studies. One small randomized controlled trial reported faster recovery in the surgery group, but this study is probably subject to selection bias as well as underpowered design. There is a need to strengthen the knowledge base regarding treatment of stress fractures in the fifth metatarsal. This study seeks to answer whether osteosynthesis with an intramedullar screw fixation gives faster painfree weight bearing compared to non-operative treatment with a walking boot.

ELIGIBILITY:
Inclusion Criteria:

* Zone 3 fracture

Exclusion Criteria:

* Neuropathy
* Open fractures
* High energy injuries
* Associated injury in the same or opposite extremity that may affect treatment or rehabilitation
* Pressure ulcer(s)
* Lack of consent competence
* Fracture radiologically confirmed more than six months ago
* No possibility of follow-up at one of the study centers
* Established pseudarthrosis
* Medical condition that contraindicates surgery
* Non-compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain free weight bearing | 2 years
  Defined as Visual Analoge Scale below 3. The scale range is 0 to 10, where 0 means "no pain" and 10 means "worst pain".

SECONDARY OUTCOMES:
Palpatory pain | 2 years
  Visual Analog Scale below 3
Radiological healing | 2 years
  Time to radiological callus formation
Work status | 2 years
  Time of sick leave
Refracture | 2 years
  Rate of refractures
Delayed union | 2 years
  Rate of delayed unions
Nonunions | 2 years
  Rate of nonunions
Level of activity | 2 years
  Time to normal activity level is resumed

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, PhD, Principal Investigator — Ostfold HT
Locations (3):
- Norway (3):
  - Østfold Hospital Trust, Grålum
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No